CLINICAL TRIAL: NCT00448071
Title: A Phase II, Randomized Double Blind Placebo-Controlled, Dose Escalating Study to Determine Pharmacokinetic and Pharmacodynamic Effects of MTR107 in End-Stage Renal Disease (ESRD) Patients
Brief Title: Pharmacokinetic and Pharmacodynamic Effects of MTR107 in End-Stage Renal Disease (ESRD) Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wolfson Medical Center (Other Government)
Collaborators: Meditor Pharmaceuticals Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MTR107IL-104
Record Dates: First submitted 2007-03-14; First posted 2007-03-15 (Estimated); Last update posted 2007-03-15 (Estimated); Status verified 2006-12

CONDITIONS: Hypotension; End Stage Renal Disease; Intra Dialytic Hypotension
Keywords: Hypotension; End Stage Renal Disease; Intra Dialytic Hypotension; ESRD; Blood Pressure; Dialysis
MeSH Terms: conditions — Hypotension; Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: MTR107

SUMMARY:
MTR107 effect on blood pressure throught the dialysis procedure and its ability to prevent Intra dialytic Hypotension

DETAILED DESCRIPTION:
The present clinical trial aims to investigate and provide a more precise characterization of the pharmacokinetic and pharmacodynamic profile of MTR107 in a population of ESRD patients predisposed to developing intradialytic hypotension. The study is also designed as a dose esclating study aiming to assess MTR107 safety.

ELIGIBILITY:
Inclusion Criteria:

1. Age 20-75 years, inclusive.
2. Presence of frequent bouts of hypotension defined as 3 or more intradialytic hypotensive events per month for the last six months prior to baseline, despite standard adjustments in dry weight.
3. ECG performed up to one month before study start.
4. Well-preserved hepatic function (within normal laboratory ranges) at study entry as judged by:

   * Serum Bilirubin (Total Bilirubin (direct and indirect) 0.3-1.0 mg/dL, and Direct Bilirubin 0.1-0.5 mg/dL)
   * Serum Albumin (>3.6 g/dL),
   * Serum aminotransferases (AST (0-37 U/L) and ALT (0-40 U/L)),
   * GGT (Gamma Glutamine Trans Peptidase)
5. Normal coagulation status at study entry as judged by PT-INR, PTT, fibrinogen and platelet count.
6. Willingness to participate in the study and adhere to the study design.
7. Willingness to sign an informed consent form.

Exclusion Criteria:

1. Uncontrolled hypertension >140/90 mmHg.
2. Unstable angina.
3. Abnormal ECG which may indicate acute disease
4. Variable weight gains.
5. Mental retardation.
6. Pregnancy.
7. Malignancy or other concomitant serious diseases.
8. Current participation in another clinical trial involving an investigational drug/device, or participation in such a trial within the last 30 days.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12
Dates: Start 2006-05; Study Completion 2007-03

PRIMARY OUTCOMES:
A descriptive pharmacokinetic / pharmacodynamic study. No primary end-points apply.

SECONDARY OUTCOMES:
Exploratory Efficacy Parameters:
 Number and type of medical interventions required for treatment of hypotension.
 Alleviation of symptoms associated with intradialytic hypotension.
 Efficiency of dialysis as reflected by Kt/V

CONTACTS AND LOCATIONS:
Overall Officials: Zeev Katzir, MD, Principal Investigator — Wolfson Medical Center; Shay Efrati, MD, Principal Investigator — Asaf Harofeh Medical Center
Locations (2):
- Israel (2):
  - Wolfson Medical Center, Holon
  - Asaf Harofeh Medical Center, Rishon LeZiyyon